CLINICAL TRIAL: NCT07105423
Title: Food Choices of the Future: The Relationship Between Mindful Eating and Sustainability in University Students
Brief Title: Mindful Eating and Sustainability
Status: Recruiting | Type: Observational
Sponsor: Atılım University (Other)
Responsible Party: Sponsor
Other Study IDs: Sedef Güngör-Atılım-01
Record Dates: First submitted 2025-05-16; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Sustainable Food Consumption; Minfullness; Mindfull Eating
Keywords: Mindfulness; Mindful eating; Sustainable eating; Sustainability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Problems such as worldwide population growth, climate change and depletion of natural resources increase the importance of sustainable nutrition. Sustainable nutrition is an approach that promotes healthy food choices, taking into account environmental, social and economic impacts. This approach affects not only the environment, but also the health of individuals and social equity. Eating mindfulness supports individuals to make both healthy and environmentally friendly choices by increasing their sensory and mental attention while eating. University students are an important target group for raising sustainability awareness as they develop independent eating habits during this period. However, it is seen that young individuals are not sufficiently informed about sustainable nutrition and eating awareness.

Aim: This study aims to examine the relationship between eating awareness and sustainable eating habits of university students.

Expected Results of the Study:

It is expected to determine the relationship between eating awareness levels and sustainable eating habits of university students. The findings are expected to show that students with high levels of eating awareness are more prone to sustainable eating habits. In addition, the links between physical activity level and sustainable nutrition will also be revealed, and it is thought that it can be concluded that physically active students are more sensitive to environmental awareness and sustainable food preferences.

DETAILED DESCRIPTION:
İntroduction:

Problems such as rapidly increasing population worldwide, climate change, depletion of natural resources and environmental degradation increase the importance of sustainable nutrition more than ever. Sustainable nutrition is defined as an approach that encourages healthy and balanced food choices by considering the environmental, social and economic impacts of food production and consumption systems. In this context, sustainability of food systems is not only limited to environmental impacts, but also has important implications for the health status of individuals and social equity.

Awareness of individuals' food choices is a critical element that directly affects both their personal health and the future of the planet. Eating mindfulness helps individuals make healthy food choices by increasing their sensory and mental attention during the eating process. This concept includes not only focusing on feelings of hunger and satiety, but also understanding the sources, nutritional values and environmental impacts of the foods eaten. Developing eating awareness can enable individuals to reduce food waste, make more informed choices regarding nutritional value, and adopt a more sustainable approach to food consumption, taking into account environmental impacts.

University students usually develop independent eating habits during this period of their lives and consider environmental, economic and health-related factors in this process. The eating habits of young people may shape their lifelong healthy eating behaviors. During this period, students' awareness of environmental awareness and sustainable food preferences becomes an important factor affecting their future food choices. However, many young individuals may not have sufficient knowledge about sustainable nutrition and eating awareness.

This study aims to examine the relationship between eating awareness and sustainable eating habits of university students. The main objectives of the project were to determine students' levels of eating awareness, their level of knowledge about sustainable food choices and the interaction between these two concepts. Based on the findings, educational programs and awareness campaigns will be proposed to promote healthy and sustainable eating habits for university students. In this context, the project aims to contribute to the adoption of healthy eating habits at both individual and societal levels.

Aim: This study aims to examine the relationship between eating awareness and sustainable eating habits of university students.

Method:

Research Design This study is based on a cross-sectional research design to examine the relationship between eating awareness and sustainable eating behaviors among university students. This design will enable the examination of the relationships between eating awareness and sustainable eating behaviors among university students.

Sample The target group of the research consists of male and female students between the ages of 18-25 years studying at universities in Ankara. The study is planned to be carried out with at least 150 participants.

Data Collection Process Participants will be informed about the purpose of the research, it will be stated that confidentiality principles will be followed, and consent will be obtained from voluntary participants. For this, individuals will fill out "Informed voluntary consent forms". Individuals who will participate in the study will be reached online or through universities. Data will be collected through online or face-to-face questionnaire applications. Participation in the study will be voluntary.

Data Collection Tools Demographic information (age, gender, height, weight, presence of chronic diseases, etc.) and information on dietary habits of the participants will be obtained with a questionnaire form.

International Physical Activity Questionnaire (IPAQ): In the study, IPAQ will be used to assess the physical activity levels of individuals. This questionnaire was developed in 1998 and designed to systematically measure the daily physical activity of individuals. The questionnaire assesses various types of physical activity (e.g., walking, light and vigorous exercise) and the weekly duration of these activities, allowing participants to determine their total physical activity level. The Turkish validity and reliability of IPAQ was performed in 2010.

Sustainable and Healthy Eating Behaviors Scale: It is a scale developed to assess individuals' behaviors towards sustainability and healthy eating habits. The adaptation, validity and reliability study of the scale into Turkish was conducted in 2023.

Eating Awareness Scale: It will be used in the study to assess individuals' levels of eating mindfulness. In the study, it will be used to assess the eating awareness levels of individuals. This scale aims to measure the quality of attention given to the eating experience in the general population as well as measuring the attention and awareness levels of individuals in the eating process. The scale aims to help individuals develop healthy eating habits by assessing emotional and mental processes related to eating experiences. The Turkish validity and reliability study of the Eating Awareness Scale was conducted in 2016. The use of the Eating Awareness Scale will be an important tool to understand the relationship between eating awareness and sustainable eating habits.

Expected Results of the Study:

It is expected to determine the relationship between eating awareness levels and sustainable eating habits of university students. The findings are expected to show that students with high levels of eating awareness are more prone to sustainable eating habits. In addition, the links between physical activity level and sustainable nutrition will also be revealed, and it is thought that it can be concluded that physically active students are more sensitive to environmental awareness and sustainable food preferences.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-25
* Volunteering
* No communication problems
* To reside in Ankara

Exclusion Criteria

* Under 18 years of age and over 25 years of age
* Those with communication problems
* Having any psychological disorder
* Not residing in Ankara

Ages: 18 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: The population of this study consisted of male and female university students aged between 18 and 25 years studying in Ankara.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
Changes in university students' mindful eating levels according to their sustainable and healthy eating behaviour scale scores | Up to two month
  The Mindful Eating Questionnaire (MEQ) will be used to assess individuals' levels of mindful eating. The 28-item, 4-point Likert-type scale has 7 sub-factors. A high score on each sub-dimension of the scale indicates that the individual possesses the trait assessed by that sub-dimension. The scale also provides a total mindful eating score. When scoring, the average of the sub-dimensions and the total score is calculated. 'Sustainable and Healthy Eating Behaviours Scale' will be used to measure sustainable eating behaviours. The scale consists of 32 questions in total and is scored on a 7-point Likert scale. The scale has a total of 7 subgroups. These are evaluated by factor scoring. Then, the total score of the scale is obtained by calculating the average of the scores obtained for 7 subgroups. The minimum value obtained from the total score is 1 and the maximum value is 7. Both subgroup and total score correlation will be analysed to determine the change between the two.

SECONDARY OUTCOMES:
Change in physical activity levels according to sustainable and healthy eating behaviour score | Up to one month
  Physical activity levels of university students will be determined using the "International Physical Activity Questionnaire (Short Form) (IPAQ-SF)". The energy required for the activities in the scale is calculated with the MET-minute score. 'Sustainable and Healthy Eating Behaviours Scale' will be used to measure sustainable eating behaviours. The scale consists of 32 questions in total and is scored on a 7-point Likert scale. The scale has a total of 7 subgroups. These are evaluated by factor scoring. Then, the total score of the scale is obtained by calculating the average of the scores obtained for 7 subgroups. The minimum value obtained from the total score is 1 and the maximum value is 7. Both subgroup and total score correlation will be analysed to determine the change between the two.
Change in physical activity levels according to mindful eating questionnaire score | Up to a month
  Physical activity levels of university students will be determined using the "International Physical Activity Questionnaire (Short Form) (IPAQ-SF)". The energy required for the activities in the scale is calculated with the MET-minute score. The Mindful Eating Questionnaire (MEQ) will be used to assess individuals' levels of mindful eating. The 28-item, 4-point Likert-type scale has 7 sub-factors. A high score on each sub-dimension of the scale indicates that the individual possesses the trait assessed by that sub-dimension. The scale also provides a total mindful eating score. When scoring, the average of the sub-dimensions and the total score is calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Köse G, Tayfur M, Birincioğlu İ. Dönmez A. Adaptation study of the Mindful Eating Questionnaire (MEQ) into Turkish. Journal of Cognitive-Behavioral Psychotherapy and Research, 2016;5(3): 125-134. doi: 10.5455/JCBPR.250644.
- [Background] Yüksel A, Yılmaz Önal H. Evaluation of University Students' Knowledge of and Practices for Sustainable Nutrition. International Journal of Agriculture Environment and Food Sciences, 2021:5(2);146-156. https://doi.org/10.31015/jaefs.2021.2.3
- [Background] Gáthy AB, Soltész AK, Szűcs I. Sustainable consumption - examining the environmental and health awareness of students at the University of Debrecen. Cogent Business & Management, 2022;9(1):2105572. https://doi.org/10.1080/23311975.2022.2105572.
- [Background] Schachtner-Appel A, Song H. A Mindful and Sustainable Eating Intervention to Improve Attitudes Related to Mindfulness, Sustainability, and Fruit and Vegetable Consumption in Elementary Schools. Journal of Human Sciences and Extension, 2024;12(1): 7. DOI: https://doi.org/10.55533/2325-5226.1447.
- [Background] Framson C, Kristal AR, Schenk JM, Littman AJ, Zeliadt S, Benitez D. Development and validation of the mindful eating questionnaire. J Am Diet Assoc. 2009 Aug;109(8):1439-44. doi: 10.1016/j.jada.2009.05.006. PMID 19631053
- [Background] Koksal E, Bilici S, Citar Daziroglu ME, Erdogan Govez N. Validity and Reliability of the Turkish Version of the Sustainable and Healthy Eating Behaviors Scale. Br J Nutr. 2022 Aug 8:1-20. doi: 10.1017/S0007114522002525. Online ahead of print. PMID 35938236
- [Background] Zakowska-Biemans S, Pieniak Z, Kostyra E, Gutkowska K. Searching for a Measure Integrating Sustainable and Healthy Eating Behaviors. Nutrients. 2019 Jan 5;11(1):95. doi: 10.3390/nu11010095. PMID 30621258
- [Background] Saglam M, Arikan H, Savci S, Inal-Ince D, Bosnak-Guclu M, Karabulut E, Tokgozoglu L. International physical activity questionnaire: reliability and validity of the Turkish version. Percept Mot Skills. 2010 Aug;111(1):278-84. doi: 10.2466/06.08.PMS.111.4.278-284. PMID 21058606
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Sogari G, Velez-Argumedo C, Gomez MI, Mora C. College Students and Eating Habits: A Study Using An Ecological Model for Healthy Behavior. Nutrients. 2018 Nov 23;10(12):1823. doi: 10.3390/nu10121823. PMID 30477101
- [Background] Nelson JB. Mindful Eating: The Art of Presence While You Eat. Diabetes Spectr. 2017 Aug;30(3):171-174. doi: 10.2337/ds17-0015. PMID 28848310
- [Background] Fanzo J, Rudie C, Sigman I, Grinspoon S, Benton TG, Brown ME, Covic N, Fitch K, Golden CD, Grace D, Hivert MF, Huybers P, Jaacks LM, Masters WA, Nisbett N, Richardson RA, Singleton CR, Webb P, Willett WC. Sustainable food systems and nutrition in the 21st century: a report from the 22nd annual Harvard Nutrition Obesity Symposium. Am J Clin Nutr. 2022 Jan 11;115(1):18-33. doi: 10.1093/ajcn/nqab315. PMID 34523669
- [Background] Fanzo J, Bellows AL, Spiker ML, Thorne-Lyman AL, Bloem MW. The importance of food systems and the environment for nutrition. Am J Clin Nutr. 2021 Jan 4;113(1):7-16. doi: 10.1093/ajcn/nqaa313. PMID 33236086